CLINICAL TRIAL: NCT00285701
Title: Early Detection of Pre-malignant and Malignant Conditions in the Colon by Means of Fluorescence Endoscopy Using Local and Oral Sensitisation With Hexaminolevulinate (HAL) - a Dose Finding Study
Brief Title: Early Detection of Polyps and Colon Cancer by Fluorescence Imaging - a Dose-finding Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCCO101/05
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

INTERVENTIONS:
Drug: hexaminolevulinate

SUMMARY:
Patients referred for colon inspection (colonoscopy) due to suspicion of colon polyps/cancer will receive local administration of hexaminolevulinate (HAL) prior to colon inspection. Blue light illumination will induce red fluorescence of polyps and tumours, improving detection of the polyps and tumors. Different HAL doses will be tested to find the optimal image conditions. Tolerability measurements will be performed to ensure patient safety.

DETAILED DESCRIPTION:
Colonoscopy is regarded as the "gold standard" for diagnosis of colorectal cancer. The sensitivity is uncertain but proposed to be (75-95%), however flat adenomas which are easily missed, are often not recognised. Fluorescence imaging may increase the sensitivity of standard white light colonoscopy by identifying more polyps and flat adenomas which will make the resection of adenomas more complete.

In this study hexaminolevulinate (HAL) will be administered locally as a photosensitiser, using different doses to find the optimal imaging conditions as well as making patient safety assessments.

Both standard white light and blue light (fluorescence) inspection will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of colorectal cancer
* Written informed consent
* Data protection consent
* 18-85 years

Exclusion Criteria:

* Liver cirrhosis
* Hepatitis
* Abnormal liver function
* Porphyria
* Patient non-compliance
* Coagulation disorder
* Contraindication to colonoscopy
* Pregnancy and lactation
* Participation in another study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Mayinger, MD, PhD, Principal Investigator — Endlicher E, et al. Hexaminolevulinate-induced fluorescence endoscopy in patients with rectal adenoma and cancer: a pilot study. Gastrointestinal Endoscopy 2004;60:449-454
Locations (1):
- Dept of Medicine, Munic-Hospital Pasing, Munich, Bavaria, Germany